CLINICAL TRIAL: NCT04712994
Title: PrEPARE: PrEP in Pregnancy, Accelerating Reach and Efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Grace John-Stewart, Associate Professor, School of Medicine: Global Health, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00008392; R01HD094630 (NIH); R01AI125498 (NIH)
Record Dates: First submitted 2020-12-30; First posted 2021-01-19 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Pre-Exposure Prophylaxis; HIV Infections; Pregnancy Related
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: A difference-in-difference design will be used; this is a quasi-experimental design that compares data before an intervention is introduced to data after the intervention is introduced and compares that with the expected change before and after in comparison clinics. One package of interventions (video-based PrEP counseling, HIV Self-Testing [HIVST], and optimized PrEP delivery) will be implemented at four intervention facilities and here will be 4 comparison facilities will undergo the same data collection procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEP Optimization Strategies (Experimental): Four facilities will be assigned to the intervention group. The intervention group will receive a pre-identified package of interventions (PrEP video counselling, HIV Self-Testing, and optimized delivery and prescription processes).
  Interventions: Other: PrEP Optimization Interventions
- Comparator (No Intervention): Four facilities will be assigned to the comparator group.

INTERVENTIONS:
Other: PrEP Optimization Interventions — A bundle of strategies (video-based PrEP counselling, HIV Self-Testing [HIVST] for women undergoing repeat HIV testing, and optimized PrEP delivery and prescription processes) will be implemented in the intervention group.
  Arms: PrEP Optimization Strategies

SUMMARY:
This study tests strategies for improving PrEP implementation in maternal and child health clinics using a difference-in-difference approach.

DETAILED DESCRIPTION:
This study aims to improve integrated delivery of PrEP to women seeking health services in maternal and child health clinics by piloting and evaluating four strategies or bundles of strategies for optimized PrEP delivery. Strategies to be tested include a pre-developed package of strategies (video counseling, HIV self-testing, and optimized delivery).

ELIGIBILITY:
Inclusion Criteria:

* Women receiving Maternal and Child Health (MCH) services HCW participating in satisfaction surveys

Exclusion Criteria:

* Unwilling or unable to provide informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Anyone presenting for maternal child health services can be included in the study.
Enrollment: 1958 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace John-Stewart, MD, MPH, PhD, Principal Investigator — University of Washington
Locations (8):
- Kenya (8):
  - Kendu Sub-District Hospital, Homa Bay
  - Ober Health Center, Homa Bay
  - Masogo Sub-County Hospital, Kisumu
  - Nyahera Sub Sub County Hospital, Kisumu
  - Bondo County Referral Hospital, Siaya
  - Madiany Sub County Hospital, Siaya
  - Malanga Health Center, Siaya
  - Uyawi Sub County Hospital, Siaya

REFERENCES:
- [Derived] Sila J, Wagner AD, Abuna F, Dettinger JC, Odhiambo B, Ngumbau N, Oketch G, Sifuna E, Gomez L, Hicks S, John-Stewart G, Kinuthia J. An implementation strategy package (video education, HIV self-testing, and co-location) improves PrEP implementation for pregnant women in antenatal care clinics in western Kenya. Front Reprod Health. 2023 Nov 17;5:1205503. doi: 10.3389/frph.2023.1205503. eCollection 2023. PMID 38045529

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrollment number in the protocol section (1958) includes the sum of participants who started in the participant flow module below (1919), as well as the 39 additional health care workers who provided cross-sectional data in the intervention group during the intervention period. There was no drop-off between consent and enrollment.
Units Other Than Participants: Facilities
Period: Baseline Period (3 Months)
Arm/Group | PrEP Optimization Strategies | Comparator
Started | 480; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.) | 480; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.)
Completed | 480; 4 Facilities | 480; 4 Facilities
Not Completed | 0; 0 Facilities | 0; 0 Facilities
Period: Intervention Period (3 Months)
Arm/Group | PrEP Optimization Strategies | Comparator
Started | 481; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.) | 479; 4 Facilities (The total population includes cross-sectional, independent groups from 2 time periods. The populations in the baseline and intervention periods are NOT expected to be the same, as they are independent, cross-sectional samples. This is a difference in differences design with 2 time periods.)
Completed | 481; 4 Facilities | 479; 4 Facilities
Not Completed | 0; 0 Facilities | 0; 0 Facilities

BASELINE CHARACTERISTICS:
Groups:
- PrEP Optimization Strategies -- Baseline; PrEP Optimization Strategies -- Intervention Period: Four facilities will be assigned to the intervention group. The intervention group will receive a pre-identified package of interventions (PrEP video counselling, HIV Self-Testing, and optimized delivery and prescription processes).
  PrEP Optimization Interventions: A bundle of strategies (video-based PrEP counselling, HIV Self-Testing [HIVST] for women undergoing repeat HIV testing, and optimized PrEP delivery and prescription processes) will be implemented in the intervention group.
- Comparator -- Baseline; Comparator -- Intervention Period: Four facilities will be assigned to the comparator group.
- Total: Total of all reporting groups
Arm/Group | PrEP Optimization Strategies -- Baseline | Comparator -- Baseline | PrEP Optimization Strategies -- Intervention Period | Comparator -- Intervention Period | Total
Number analyzed (Participants) | 480 | 480 | 481 | 479 | 1920
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [21 to 29] | 25 [21 to 30] | 25 [22 to 30] | 25 [22 to 30] | 25 [21 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 480 | 480 | 481 | 479 | 1920
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 480 | 480 | 481 | 479 | 1920
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 480 | 480 | 481 | 479 | 960

OUTCOME MEASURES:

1. Primary Outcome: PrEP Penetration
Description: Proportion of women who are screened for PrEP / total women receiving antenatal or postnatal services
Time Frame: 6 months
Population: The total population includes cross sectional groups from 2 time periods. The population analyzed above is a summation of the participants analyzed in the 2 periods. This is a difference in differences design with 2 time periods.
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP Optimization Strategies | Comparator
Number analyzed (Participants) | 961 | 958
Participants
  Baseline: number analyzed (Participants) | 480 | 480
  Baseline | 30 | 17
  Intervention: number analyzed (Participants) | 481 | 478
  Intervention | 46 | 8

2. Primary Outcome: PrEP Fidelity
Description: Proportion of women who receive all PrEP specific steps in a visit: HIV testing, HIV risk screening, PrEP counseling
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP Optimization Strategies | Comparator
Number analyzed (Participants) | 961 | 958
Participants
  Baseline: number analyzed (Participants) | 480 | 480
  Baseline | 14 | 4
  Intervention: number analyzed (Participants) | 481 | 478
  Intervention | 28 | 5

3. Primary Outcome: Timeliness of Services
Description: Time (minutes) spent receiving services from health care works
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | PrEP Optimization Strategies | Comparator
Number analyzed (Participants) | 384 | 384
minutes
  Baseline: number analyzed (Participants) | 192 | 192
  Baseline | 18 [12 to 36] | 16 [10 to 33]
  Intervention: number analyzed (Participants) | 192 | 192
  Intervention | 17 [11 to 29] | 14 [9 to 27.5]

4. Primary Outcome: Waiting Time
Description: Time (minutes) spent waiting to receive services
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | PrEP Optimization Strategies | Comparator
Number analyzed (Participants) | 384 | 384
minutes
  Baseline: number analyzed (Participants) | 192 | 192
  Baseline | 49 [22.5 to 77] | 37 [14.5 to 74]
  Intervention: number analyzed (Participants) | 192 | 192
  Intervention | 55 [31 to 80] | 29 [14 to 46.5]

5. Primary Outcome: HCW Acceptability
Description: Total on 4 item Acceptability of Intervention Measures (AIM) score, 1 (Completely disagree) to 5 (Completely Agree) Likert scale. The minimum score on the 4 items is 4 points (scoring 1 on each of the 4 items) while the maximum is 20 points (scoring 5 on each of the 4 items). A higher score indicates a better outcome. The sub-scores on each of the 4 items are summed.
Time Frame: 6 months
Population: This outcome was assessed on a group of 39 HCW who were involved in delivering the implementation strategy package. These are not a subset of the women enrolled in the study, hence the numbers are not concordant.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PrEP Optimization Strategies
Number analyzed (Participants) | 39
score on a scale | 20.0 [16.0 to 20.0]

6. Primary Outcome: Health Care Worker (HCW) Appropriateness
Description: Total on 4 item Intervention Appropriateness Measure (IAM) score, 1 (Completely disagree) to 5 (Completely Agree) Likert scale. The minimum score on the 4 items is 4 points (scoring 1 on each of the 4 items) while the maximum is 20 points (scoring 5 on each of the 4 items). A higher score indicates a better outcome. The sub-scores on each of the 4 items are summed.
Time Frame: 6 months
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PrEP Optimization Strategies
Number analyzed (Participants) | 39
score on a scale | 19.5 [16.0 to 20.0]

7. Primary Outcome: Client Satisfaction
Description: Total on 6 item exit survey of clients to assess their satisfaction with services received at the facility, 1 (worse) to 4 (better) scale. The minimum score on the 6 items is 6 points (scoring 1 on each of the 6 items) while the maximum is 24 points (scoring 4 on each of the 6 items). A higher score indicates a better outcome. The sub-scores on each of the 4 items are summed.
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PrEP Optimization Strategies | Comparator
Number analyzed (Participants) | 961 | 958
score on a scale
  Baseline: number analyzed (Participants) | 480 | 480
  Baseline | 21.0 [19.0 to 23.0] | 23.0 [20.0 to 23.0]
  Intervention: number analyzed (Participants) | 481 | 478
  Intervention | 23.0 [21.0 to 23.0] | 23.0 [20.0 to 24.0]

8. Secondary Outcome: PrEP Uptake
Description: Proportion of women who accept PrEP among those offered
Time Frame: 6 months
Population: The total population includes cross sectional groups from 2 time periods. The population analyzed above is a summation of the participants analyzed in the 2 periods. This is a difference in differences design with 2 time periods.
  This analysis population is a subset of the total because it only includes those who were offered PrEP, as noted in the denominator description of the indicator.
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP Optimization Strategies | Comparator
Number analyzed (Participants) | 34 | 17
Participants
  Baseline: number analyzed (Participants) | 6 | 8
  Baseline | 0 | 1
  Intervention: number analyzed (Participants) | 28 | 9
  Intervention | 0 | 1

9. Secondary Outcome: PrEP Continuation
Description: Proportion of women who present for a refill among those initially prescribed PrEP
Time Frame: 6 months
Population: The total population includes cross sectional groups from 2 time periods. The population analyzed above is a summation of the participants analyzed in the 2 periods. This is a difference in differences design with 2 time periods.
  This analysis population is a subset of the total because it only includes those who were initially prescribed PrEP, as noted in the denominator description of the indicator.
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP Optimization Strategies | Comparator
Number analyzed (Participants) | 36 | 17
Participants
  Baseline: number analyzed (Participants) | 8 | 8
  Baseline | 1 | 1
  Intervention: number analyzed (Participants) | 28 | 9
  Intervention | 1 | 2

10. Secondary Outcome: PrEP Adherence
Description: Proportion of women who have >80 percent adherence to PrEP by pill count among those initially prescribed PrEP
Time Frame: 6 months
Population: During preparatory activities for data collection, it was determined that it was not feasible to extract patient adherence information; this outcome was neither collected nor compared.
Arm/Group | PrEP Optimization Strategies | Comparator
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: PrEP Efficiency
Description: Patient flow mapping to identify more efficient client flows with fewer transitions between physical spaces and providers
Time Frame: 6 months
Population: During preparatory activities for data collection, it was determined that it was not feasible to collect efficiency this outcome was neither collected nor compared.
Arm/Group | PrEP Optimization Strategies | Comparator
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Client PrEP Knowledge
Description: Number of participants with perfect knowledge on PrEP information questions based on content covered in counseling sessions
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP Optimization Strategies | Comparator
Number analyzed (Participants) | 961 | 958
Participants
  Baseline: number analyzed (Participants) | 480 | 480
  Baseline | 5 | 0
  Intervention: number analyzed (Participants) | 481 | 478
  Intervention | 56 | 5

ADVERSE EVENTS:
Time Frame: 1 cross-sectional visit. In this cross-sectional study, there were no participants followed longitudinally. Adverse events were not collected systematically within this minimal risk, cross-sectional study.
Description: We have revised the Participant Flow module, which should now allow these numbers to be consistent.
Arm/Group | PrEP Optimization Strategies | Comparator
All-Cause Mortality (participants affected / at risk) | 0/961 | 0/958
Serious Adverse Events (participants affected / at risk) | 0/961 | 0/958
Other Adverse Events (participants affected / at risk) | 0/961 | 0/961

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT04712994/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT04712994/ICF_001.pdf